CLINICAL TRIAL: NCT05939050
Title: The Long-term Effect on Oral Health Using a Powered Toothbrush in Individuals With Mild Cognitive Impairment: An Intervention Trial
Brief Title: The Long-term Effect on Oral Health Using a Powered Toothbrush in Individuals With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Blekinge Institute of Technology (Other)
Collaborators: Kristianstad University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BTH-6.1.1-0085-2023
Record Dates: First submitted 2023-06-13; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Oral Health; Quality of Life
Keywords: Mild Cognitive Impairment; Oral Health; Quality of Life; Powered toothbrush
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Partisipants (Experimental)
  Interventions: Device: Powered toothbrush

INTERVENTIONS:
Device: Powered toothbrush — Oral-B Powered toothbrush

SUMMARY:
For this study, 213 individuals with Mild Cognitive Impairment were recruited. The study period ran from June 2018 to October 2021. The procedure involved a combined screening and baseline examination, including oral, medical, cognitive, and quality-of-life examinations. Re-examinations followed this at 6, 12, and 24 months. The examinations were performed at a university research clinic, and all participants received their usual medical and dental care during the study. At baseline, each participant received a powered toothbrush. Participants were carefully instructed on how to operate the powered toothbrush and were asked to brush for at least two minutes in the morning and evening. No restrictions were given against the use of other oral care products. Compliance with the powered toothbrush was followed by a participant survey conducted at each examination.. Facilitating and improving life by introducing a powered toothbrush as part of oral hygiene may benefit individuals with MCI. This study aimed to investigate whether the use of a powered toothbrush could maintain or improve oral health by reducing dental plaque (PI), bleeding on probing (BOP), and periodontal pocket depth (PPD)≥4mm in a group of individuals with MCI for an observation period of 24 months. Furthermore, to study how oral health changes affect QoL aspects.

ELIGIBILITY:
Inclusion Criteria:

* Being 55 years or older
* Having experienced memory problems in the last six months before inclusion
* Having a Mini-Mental State Examination score of 20-28
* Are not receiving any formal care
* Having at least ten teeth of their own

Exclusion Criteria:

* Having a terminal illness with less than three years of expected survival
* Having another known significant cause of disease explaining cognitive impairment

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Change in the amount of dental plaque | From baseline, to month 6, and to month 12, and to month 24, and to month 36
  Presence of dental plaque measured on four of the tooth surfaces presented as a percentage
Change in the amount of gingival bleeding on probing | From baseline, to month 6, and to month 12, and to month 24, and to month 36
  Number of bleeding from the gingiva measured on four sides of the teeth presented as a percentage
Change in the number of periodontal pockets 4 mm or deeper | From baseline, to month 6, and to month 12, and to month 24, and to month 36
  The number of periodontal pockets 4 mm or deeper measured on four of the tooth surfaces presented as a percentage
Change in values for the quality of life instrument QoL-AD | From baseline, to month 6, and to month 12, and to month 24, and to month 36
  The value for the quality of life instrument QoL-AD (Quality of Life Alzheimer Disease) is measured on a scale from 0-30, where 30 corresponds to the highest quality of life
Change in values for the oral health related quality of life instrument OHIP-14 | From baseline, to month 6, and to month 12, and to month 24, and to month 36
  The value for the oral health-related quality of life instrument OHIP-14 (Oral Health Impact Profile-14) is measured on a scale from 0-56 where 0 corresponds to the highest quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Johan Sanmartin-Berglund, Professor, Study Chair — Blekinge Institute of Technology
Locations (2):
- Sweden (2):
  - Blekinge Institute of Technology, Karlskrona
  - Johan Flyborg, Karlskrona

IPD SHARING:
Plan to Share IPD: Yes
The trial protocol and the datasets used and analyzed during the current study are available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Available after publication
Access Criteria: Available from the corresponding author upon reasonable request.

REFERENCES:
- [Derived] Flyborg J, Renvert S, Anderberg P, Sanmartin-Berglund J. The long-term effect on oral health and quality of life using a powered toothbrush in individuals with mild cognitive impairment. An intervention trial. Spec Care Dentist. 2024 Nov-Dec;44(6):1700-1708. doi: 10.1111/scd.13040. Epub 2024 Jul 12. PMID 38994574